CLINICAL TRIAL: NCT06807307
Title: KEAPnes: Transcriptional Framework for the Molecular Diagnosis of Response to Immunotherapy in Lung Cancer With Agnostic Potential
Brief Title: Transcriptional Framework for the Molecular Diagnosis of Response to Immunotherapy in Lung Cancer With Agnostic Potential
Acronym: KEAPnes
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS158/IRE/24
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: NSCLC

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective court of identification: The retrospective identification cohort consists of patients with metastatic disease treated with front line immunotherapy as per clinical practice from 2017 to 2021 at the IRCCS National Cancer Institute "Regina Elena".
  The optimal parameters for identifying KEAPness and obtaining information on the interactions between pairs of genes fundamental for the activation of KEAPness itself.
- Prospective validation cohort: The validation court will collect NSCLC patients (metastatic setting, treated with first-line immunotherapy possibly in association with chemotherapy as per clinical practice) and also pancancer patients (patients with metastatic cancer other than NSCLC and who have received an ICI, either alone or in association with other medical treatments as per clinical practice), from which patients with NSCLC are excluded (PCC cohort). These patients will be recruited from the collaborating institute IRCCS Pascale of Naples. To ensure reproducibility of the study, the same approach of the first court will be applied to this one, i.e. the optimal parameters will be set for the identification of KEAPness and to obtain information on the interactions between pairs of genes fundamental for the activation of KEAPness.

SUMMARY:
Through genomic and transcriptomic sequencing techniques (whole exome sequencing, WES; whole transcriptome sequencing, WTS) patients with enrichment for KEAPness and specific gene interactions associated with it.

DETAILED DESCRIPTION:
Retrospective-prospective, non-pharmacological, biological, multicenter observational study, for which the collection and use of tissue samples from patients suffering from NSCLC and/or other tumor types. Through genomic and transcriptomic sequencing techniques (whole exome sequencing, WES; whole transcriptome sequencing, WTS) patients with enrichment for KEAPness and specific gene interactions associated with it. Subsequently, through the same techniques, applied to different tumor regions taken from operating site it will be possible to identify the evolution of the tumor at a spatio-temporal level and the immune subtype associated with the presence/absence of KEAPness. Finally, cell lines will be used to recapitulate what was observed in the patient and per-patient cohorts identify new pharmacological vulnerabilities associated with the characteristics of KEAPness.

ELIGIBILITY:
Inclusion Criteria cohort (NSCLC-IC):

* Age >18 years;
* Histological diagnosis of NSCLC
* metastatic disease
* Availability, at the time of enrollment, of adequate biological material to be able to perform molecular analyses, taken (surgical or by biopsy) before administration of any anti-tumor treatment (chemotherapy and/or radiotherapy);
* ECOG PS 0-2;
* Adequate hematological, hepatic and renal function;
* Measurable disease according to RECIST criteria
* Availability of follow-up data for at least 6 months and/or until death/progression

Exclusion Criteria cohort (NSCLC-IC):

* Previous systemic therapy for metastatic disease;
* Comorbidities not controlled with adequate medical therapy.

Inclusion Criteria NSCLC-VC cohort:

* Age >18 years;
* Histological diagnosis of NSCLC
* metastatic disease
* Availability, at the time of enrollment, of adequate biological material to be able to perform molecular analyses, taken (during surgery and/or by biopsy) before administration of any anti-tumor treatment (chemotherapy and/or radiotherapy);
* ECOG PS 0-2;
* Adequate hematological, hepatic and renal function;
* Measurable disease according to RECIST criteria;
* Written informed consent (participation in the study and data processing)

Exclusion Criteria NSCLC-VC cohort:

* Previous systemic treatment for metastatic disease;
* Comorbidities not controlled with adequate medical therapy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic NSCLC who are candidates for and/or undergoing treatment first-line chemotherapy-immunotherapy combination treatment or immunotherapy from alone (if PD-L1>50% as per clinical practice) that meet the following criteria.
Sampling Method: Non-Probability Sample
Enrollment: 256 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-06-04 (Estimated); Study Completion 2026-06-04 (Estimated)

PRIMARY OUTCOMES:
Innovative molecular tool | 24 months
  To generate an innovative molecular tool for prediction DNA/RNA will be extracted from 5μm FFPE tissue sections using the AllPrep DNA/RNA FFPE kit (Qiagen). The quality of the RNA will be evaluated with the Bioanalyzer, the integrity of genomic DNA through the Agilent NGS FFPE qPCR QC Kit (Agilent). The libraries for RNA-Seq will be prepared using the RNA TruSeq Exome Kit (Illumina). The quality of the libraries resulting will be checked using Bioanalyzer (high sensitivity DNA kit). The intermediate library before exon enrichment will be quantified with Qubit, the final library with qPCR. The samples will be sequenced in paired-end mode, sequencing 76 bp on each side. The Exome DNA sequencing will be performed using SureSelectXT Low Input Kit reagents for the initial preparation of the library followed by enrichment with Clinical Research Exome Kit (Agilent).

SECONDARY OUTCOMES:
Tracing the evolutionary path | 24 months
  Tracing the evolutionary path of NRF-2 dependent tumors, in his association with the microenvironment, and in particular the related immune subtypes, and characterize the interactions between pairs of genes (epistatic) underlying the KEAPness.i phenotype, the multi-region sequencing technology that will be used involves the use of surgical samples, taken in a single session. This allows you to isolate different regions of the tumor, corresponding to different time points (central region, R1; expansion zone, R2; locoregional metastases, R3).
  Through this methodology it is possible to trace the evolution of the tumor over time, and in particular the interactions between pairs of mutant genes linked to the KEAPness phenotype.
Identification of therapeutic vulnerabilities specific | 24 months
  Identification of therapeutic vulnerabilities specific to biological processes related to KEAPness. Cell lines derived from patients affected by NSCLC and GC, already available in the laboratories of Promoter/IFO, will initially be characterized by genomic sequencing and transcriptomic (WES and WTS) to identify the enrichment in the KEAPness phenotype and previously identified epistatic interactions.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS National Cancer Institute "Regina Elena", Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided